CLINICAL TRIAL: NCT00093496
Title: A Phase II Trial Of Gemcitabine in Combination With 17-Allylaminogeldamycin (17-AAG) In Advanced Epithelial Ovarian And Primary Peritoneal Carcinoma
Brief Title: Gemcitabine Hydrochloride and Tanespimycin in Treating Patients With Recurrent Advanced Ovarian Epithelial or Peritoneal Cavity Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00052; NCI-2009-00052 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000388036; NCI-6307; MAYO-MC0362; MC0362 (Other: Mayo Clinic); 6307 (Other: CTEP); P30CA015083 (NIH); N01CM62205 (NIH); NCT01646918 (obsolete NCT alias); NCT01664312 (obsolete NCT alias)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2011-10

CONDITIONS: Primary Peritoneal Cavity Cancer; Recurrent Ovarian Epithelial Cancer; Stage III Ovarian Epithelial Cancer; Stage IV Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Gemcitabine; tanespimycin

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients are stratified according to gemcitabine hydrochloride therapy (gemcitabine hydrochloride-naive/no prior exposure to gemcitabine hydrochloride vs gemcitabine hydrochloride-resistant/prior exposure to gemcitabine hydrochloride as a single agent with disease progression while on treatment). Patients receive tanespimycin IV over 2 hours on days 1 and 8 during course 1 and days 2 and 9 during subsequent courses and gemcitabine hydrochloride IV over 30 minutes on day 7 during course 1 and days 1 and 8 during subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.
  Interventions: Drug: gemcitabine hydrochloride; Drug: tanespimycin

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: tanespimycin — Given IV
  Other Names: 17-AAG

SUMMARY:
Phase II trial to study the effectiveness of gemcitabine hydrochloride and tanespimycin in treating patients who have recurrent advanced ovarian epithelial or primary peritoneal cavity cancer. Drugs used in chemotherapy, such as gemcitabine hydrochloride and tanespimycin, work in different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate, time to progression, and survival of patients with recurrent advanced ovarian epithelial or primary peritoneal cavity cancer treated with gemcitabine hydrochloride and 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) (tanespimycin).

II. Determine the toxicity of this regimen in these patients. III. Correlate the effect of 17-AAG alone on chaperone and client proteins in tumor samples and peripheral blood mononuclear cells with response, time to progression, and survival of these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to gemcitabine hydrochloride therapy (gemcitabine hydrochloride-naive/no prior exposure to gemcitabine hydrochloride vs gemcitabine hydrochloride-resistant/prior exposure to gemcitabine hydrochloride as a single agent with disease progression while on treatment). Patients receive tanespimycin intravenously (IV) over 2 hours on days 1 and 8 during course 1 and days 2 and 9 during subsequent courses and gemcitabine hydrochloride IV over 30 minutes on day 7 during course 1 and days 1 and 8 during subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ovarian epithelial or primary peritoneal cavity cancer

  * Relapsed disease
  * Persistent disease
* Platinum-resistant disease, defined as having evidence of disease that would be expected to be non-responsive to additional platinum-containing regimens or contraindication to platinum-based chemotherapy and 1 of the following:

  * Failure to obtain a complete response to initial platinum therapy
  * Recurrence < 6 months after completing a platinum-containing regimen for initial or recurrent disease
  * Any of the above situations and following treatment with additional chemotherapy regimens (e.g., non-platinum containing regimens)
  * Relative or absolute contraindication to platinum-based chemotherapy regimens (e.g., platinum allergy) as determine by the investigator
* Measurable or evaluable disease

  * Patients with a rising CA 125 level, even in the absence of other indicators of disease, allowed provided CA 125 is ≥ 2 times upper limit of normal (ULN)
* Patients with accessible disease must be willing to undergo tumor biopsies
* No CNS metastases
* Performance status - ECOG 0-2
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL
* Bilirubin normal
* Alkaline phosphatase ≤ 2.5 times ULN
* AST ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Ejection fraction > 40% by ECHO for patients with prior anthracycline therapy
* No significant cardiac disease including any of the following:

  * New York Heart Association class III or IV heart disease
  * History of myocardial infraction within the past year
  * Uncontrolled dysrhythmias or requirement for antiarrhythmic drugs
  * Poorly controlled angina
* No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No history of QTc ≥ 500 msec
* No active ischemic heart disease within the past 12 months
* No congenital long QT syndrome
* No left bundle branch block
* No cardiac symptoms ≥ grade 2
* No history of cardiac toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone, bleomycin, or carmustine)
* Does not meet the medicare criteria for home oxygen
* No pulse oximetry at rest and exercise < 88%
* No symptomatic pulmonary disease requiring medication including any of the following:

  * Dyspnea on or off exertion
  * Paroxysmal nocturnal dyspnea
  * Oxygen requirement
  * Significant pulmonary disease (e.g., chronic obstructive/restrictive pulmonary disease)
* No pulmonary symptoms ≥ grade 2
* No history of pulmonary toxicity after receiving anthracyclines (e.g., doxorubicin hydrochloride, daunorubicin hydrochloride, mitoxantrone, bleomycin, or carmustine)
* K+, Mg ++, and Ca ++ normal
* No seizure disorder
* No uncontrolled infection
* No history of serious allergic reaction to eggs
* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior biologic therapy
* No concurrent immunotherapy
* No concurrent routine or prophylactic colony-stimulating factors (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])
* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered
* Prior gemcitabine hydrochloride allowed provided 1 of the following criteria is met:

  * Patients have no prior exposure to gemcitabine hydrochloride
  * Patients who have prior exposure to gemcitabine hydrochloride as a single agent have experienced progressive disease while on treatment
* No other concurrent chemotherapy
* No prior radiotherapy to > 25% of bone marrow
* No history of radiotherapy that potentially included the heart in the field (e.g., mantle)

  * Chest wall irradiation or other radiotherapy techniques that do not include the heart in the radiation field area allowed
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior radiopharmaceuticals
* No concurrent radiotherapy
* No other concurrent investigational therapy
* No concurrent medications that may prolong QTc

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-10; Primary Completion 2010-04 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Haluska, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-nine patients were enrolled between November 15, 2007 and October 29, 2009. Two participants were found to be ineligible and two participants had major protocol violations. Therefore, we summarize baseline characteristics and adverse events using all 29 patients, but report endpoint analyses using 25 participants.
Pre-assignment Details: Participants were divided into two groups according to their prior gemcitabine exposure. Cohort 1 participants had no prior exposure to gemcitabine. Cohort 2 was comprised of participants with prior exposure to gemcitabine as a single agent or had experienced disease progression while on gemcitabine therapy.
Groups:
- Cohort 1 (No Prior Gemcitabine Exposure): Patients with no prior gemcitabine exposure receive tanespimycin IV over 2 hours on days 1 and 8 during course 1 and days 2 and 9 during subsequent courses and gemcitabine hydrochloride IV over 30 minutes on day 7 during course 1 and days 1 and 8 during subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.
- Cohort 2 (Prior Gemcitabine Exposure): Patients with prior gemcitabine exposure receive tanespimycin IV over 2 hours on days 1 and 8 during course 1 and days 2 and 9 during subsequent courses and gemcitabine hydrochloride IV over 30 minutes on day 7 during course 1 and days 1 and 8 during subsequent courses. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.
Period: Overall Study
Arm/Group | Cohort 1 (No Prior Gemcitabine Exposure) | Cohort 2 (Prior Gemcitabine Exposure)
Started | 15 | 14
Completed | 14 | 11
Not Completed | 1 | 3
Not completed — Protocol Violation | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (No Prior Gemcitabine Exposure) | Cohort 2 (Prior Gemcitabine Exposure) | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Median (Full Range); unit: years] | 64 [28 to 79] | 63.5 [51 to 87] | 64 [28 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Experience a Confirmed Response According to Modified RECIST Criteria.
Description: Objective response will be measured using the modified RECIST criteria. A confirmed response requires an objective status of complete or partial response on 2 consecutive evaluations occurring 4 or more weeks apart.
  Complete Response (CR): Disappearance of all target lesions and normalization of tumor biomarkers.
  Partial Response (PR): At least a 30% decrease in the sum of the target lesions from the baseline.
Time Frame: Participants were evaluated every 6 weeks on treatment, with median treatment length of 12 weeks (3 week minimum and 42 week maximum).
Population: In Cohort 1, one patient was found to be ineligible. In Cohort 2, one patient was ineligible and two patients had protocol violations. Therefore, 14 participants in Cohort 1 and eleven participants in Cohort 2 were analyzed for the primary endpoint.
Measure: Number; unit: proportion of participants
Arm/Group | Cohort 1 (No Prior Gemcitabine Exposure) | Cohort 2 (Prior Gemcitabine Exposure)
Number analyzed (Participants) | 14 | 11
proportion of participants
  Confirmed Partial Response (PR) | 0.071 | 0
  Confirmed Complete Response (CR) | 0 | 0

2. Secondary Outcome: Times to Progression
Description: Defined as the time from registration to the date of progression or last follow-up, whichever comes first. Estimated using the method of Kaplan-Meier
Time Frame: Participants were evaluated every 6 weeks on treatment (maximum 42 weeks), and followed up to 5 years from registration.
Population: An interim analysis was done on the first 12 eligible participants in each cohort. Due to drug shortage and lack of clinical activity, the interim analysis for Cohort 2 was conducted on the first 11 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (No Prior Gemcitabine Exposure) | Cohort 2 (Prior Gemcitabine Exposure)
Number analyzed (Participants) | 12 | 11
months | 1.6 [1.2 to 3.5] | 2.7 [1.3 to 5.1]

3. Secondary Outcome: Overall Survival
Description: Defined as the time from registration to date of last follow-up or death due to any cause. Estimated using the method of Kaplan-Meier.
Time Frame: Every 3 months until disease progression and then every 6 months for up to 5 years.
Population: An interim analysis was done on the first 12 eligible participants in each cohort. Due to drug shortage and lack of clinical acttivity, the interim analysis for Cohort 2 was conducted on the first 11 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1 (No Prior Gemcitabine Exposure) | Cohort 2 (Prior Gemcitabine Exposure)
Number analyzed (Participants) | 12 | 11
months | 18.3 [6.2 to NA] — There was not a sufficient number of events to estimate the upper 95% confidency level. | 11.5 [4.0 to 13.7]

4. Secondary Outcome: Toxicity
Description: Defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 as an adverse event classified as either possibly, probably, or definitely related to study treatment. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Time Frame: Participants were evaluated every 6 weeks on treatment (maximum 42 weeks)
Population: In Cohort 1, one patient was found to be ineligible. In Cohort 2, one patient was ineligible and two patients had protocol violations. Therefore, 14 participants in Cohort 1 and eleven participants in Cohort 2 were analyzed for adverse events.
Measure: Number; unit: events
Arm/Group | Cohort 1 (No Prior Gemcitabine Exposure) | Cohort 2 (Prior Gemcitabine Exposure)
Number analyzed (Participants) | 14 | 11
events
  Grade 3 | 9 | 7
  Grade 4 or Higher | 0 | 0

ADVERSE EVENTS:
Groups:
- All Patients Receiving Gemcitabine: All patients receiving gemcitabine were combined to analyze toxicity.
Arm/Group | All Patients Receiving Gemcitabine
Serious Adverse Events (participants affected / at risk) | 10/29
Other Adverse Events (participants affected / at risk) | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Receiving Gemcitabine (N=29)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (5)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Edema limbs (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (5)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Receiving Gemcitabine (N=29)
Hemoglobin decreased (Blood and lymphatic system disorders) | 24 (79)
Abdominal pain (Gastrointestinal disorders) | 3 (6)
Constipation (Gastrointestinal disorders) | 3 (8)
Diarrhea (Gastrointestinal disorders) | 9 (15)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 16 (26)
Stomach pain (Gastrointestinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 10 (13)
Edema limbs (General disorders) | 1 (3)
Fatigue (General disorders) | 7 (19)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Alkaline phosphatase increased (Investigations) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 8 (12)
Leukocyte count decreased (Investigations) | 14 (29)
Neutrophil count decreased (Investigations) | 17 (33)
Platelet count decreased (Investigations) | 9 (22)
Anorexia (Metabolism and nutrition disorders) | 4 (9)
Dizziness (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (15)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (10)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less